CLINICAL TRIAL: NCT02180152
Title: Postprandial Walking in Obese Pregnant Women and Perinatal Outcomes - a Multicenter Randomized Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, João Guilherme Bezerra Alves, PhD, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Caminhadas2014
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Gestational Diabetes; Preeclampsia
Keywords: Perinatal outcomes
MeSH Terms: conditions — Obesity; Diabetes, Gestational; Pre-Eclampsia

ARMS (2):
- Postprandial walk (Experimental)
  Interventions: Behavioral: Postprandial walks
- sedentary pregnant women (No Intervention)

INTERVENTIONS:
Behavioral: Postprandial walks — Obese pregnant women will be target to carry out walks lasting 10' after the main meals (breakfast, lunch and dinner), Monday to Friday, during 8 weeks. Adherence to the program will be determined by daily readings of pedometers previously provided to pregnant women; minimum of 1500 steps per day from Monday to Friday.
  Arms: Postprandial walk

SUMMARY:
The purpose of this study is to verify if postprandial walks are effective in obese pregnant women, as regards to gestational weight gain and typical diseases of that period, as gestational diabetes and preeclampsia. Perinatal outcomes will be observed, such as macrosomia, shoulder dystocia and fetal death.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years;
* Gestational age ≤ 20 weeks, calculated from the last menstrual period and confirmed by the first ultrasound scan;
* Obesity - body mass index ( BMI ) ≥ 30 kg/m2, based on the weight before pregnancy, reported by pregnant women no more than 5 kg below measured at admission to the study;
* Physically inactive - according to the International Physical Activity Questionnaire (IPAC);
* Single pregnancy.

Exclusion Criteria:

* Kidney disease or collagen;
* Previous history of GDM;
* Diabetes type 1 or type 2;
* Hypertensive disorders related to pregnancy;
* Hemodynamic instability;
* Vaginal bleeding;
* Visual, auditory or cognitive impairment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Weight gain after postprandial walks in obese pregnant women. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joao GB Alves, PhD, Study Director — Instituto de Medicina Integral Professor Fernando Figueira; Isabelle EA Pontes, Master, Principal Investigator — Instituto de Medicina Integral Prof. Fernando Figueira
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- See also: Click here for more informations about the Instituto de Medicina Integral Professor Fernando Figueira — http://www.imip.org.br